CLINICAL TRIAL: NCT03172156
Title: Multicentre, Prospective, Open Clinical Study of Postoperative ctDNA Dynamic Monitoring and Its Role of Prognosis in Patients With Stage I Non-small Cell Lung Cancer (NSCLC) Using Secondary Gene Sequencing (NGS)
Brief Title: ctDNA Dynamic Monitoring and Its Role of Prognosis in Stage I NSCLS by NGS
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, professor, Sun Yat-sen University
Other Study IDs: GASTO1018
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer Stage I
Keywords: NSCLC; stage I; The next generation of high-throughput gene sequencing (NGS); ctDNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA of stage I non-small cell lung cancer (NSCLC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage I NSCLC patients after surgery with ctDNA detection: Stage I NSCLC patients;ctDNA detection
  Interventions: Genetic: ctDNA detection

INTERVENTIONS:
Genetic: ctDNA detection — To detect ctDNA in Patients With Stage I Non-small Cell Lung Cancer (NSCLC) Using Secondary Gene Sequencing (NGS)

SUMMARY:
CtDNA detection is a noninvasive detection method, and the second generation of high-throughput gene sequencing (NGS) is an important means of detecting ctDNA, which can detect trace ctDNA from smaller plasma samples. This project is to study the role of ctDNA dynamic monitoring of stage I NSCLC by NGS technique to verify the prognostic predictive effect of ctDNA .

DETAILED DESCRIPTION:
CtDNA detection as a noninvasive detection method, can truly reflect the real tumor tissue gene mutation map and frequency, is the evaluation of therapeutic effect and the important monitoring indicators of clinical follow-up after treatment. The second generation of high-throughput gene sequencing (NGS) is an important means of detecting ctDNA, which can detect trace ctDNA from smaller plasma samples. The ctDNA dynamic monitoring of stage I non-small cell lung cancer (NSCLC) was performed by the second generation gene sequencing (NGS) technique to verify the prognostic predictive effect of ctDNA in stage I NSCLC patients without radiotherapy and targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative histopathological diagnosis of TNM stage IA / IB NSCLC with R0 resection;
* No adjuvant chemotherapy, radiotherapy, targeted drug therapy or biotherapy after surgery;

General selection criteria:

* Men or women of age ≥18 years and <75 years old;
* ECOG behavior status score 0 to 1;

Exclusion Criteria:

* Patients with other cancers other than NSCLC within five years prior to this study;
* who can not get enough tumor histological specimens (non-cytological) for analysis;
* human immunodeficiency virus (HIV) infection;
* NSCLC mixed with patients with small cell lung cancer;
* pregnant or lactating women;
* There is a clear history of neurological or mental disorders, including epilepsy or dementia;
* Conditions that investigators think is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Stage I Non-small Cell Lung Cancer (NSCLC) without Postoperative radiotherapy and chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years after the last patient enrolled
  Disease-free survival was assessed from surgery to disease recurrence or death as a result of any cause

SECONDARY OUTCOMES:
Overall survival | 5 years after the last patient enrolled
  Overall survival was assessed from surgery to death as a result of any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Si-Yu Wang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will not share IPD to other researchers until initial experimental conclusions is reached.

REFERENCES:
- [Derived] Yang W, You N, Jia M, Yeung SJ, Ou W, Yu M, Wang Y, Fu X, Zhang Z, Yang J, Lao Z, Liu Z, Zeng B, Ou Q, Wu X, Shao YW, Hong X, Wang S, Cheng C. Undetectable circulating tumor DNA levels correlate with low risk of recurrence/metastasis in postoperative pathologic stage I lung adenocarcinoma patients. Lung Cancer. 2020 Aug;146:327-334. doi: 10.1016/j.lungcan.2020.06.009. Epub 2020 Jun 20. PMID 32623075